CLINICAL TRIAL: NCT06297044
Title: Neural and Cognitive Correlates of Pragmatic Communication Abilities
Brief Title: Neural and Cognitive Correlates of Pragmatic Abilities
Acronym: APACS_Neuro
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 2017.20
Record Dates: First submitted 2024-02-05; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Right Hemispheric Stroke; Left Hemispheric Stroke; Traumatic Brain Injury; Right Hemispheric Brain Tumor; Left Hemispheric Brain Tumor; Mild Cognitive Impairment; Healthy
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Right Hemispheric Stroke: Specific inclusion criteria for this participants' group are:
  - unilateral right hemispheric lesion after an ischemic or hemorrhagic stroke.
  There are no specific exclusion criteria for this participants' group (see general exclusion criteria).
  Participants will undergo a detailed neuropsychological assessment as detailed in the study's detailed description and outcome measures sections.
  Interventions: Other: Neuropsychological assessment
- Left Hemispheric Stroke: Specific inclusion criteria for this participants' group are:
  - unilateral left hemispheric lesion after an ischemic or hemorrhagic stroke.
  There are no specific exclusion criteria for this participants' group (see general exclusion criteria).
  Participants will undergo a detailed neuropsychological assessment as detailed in the study's detailed description and outcome measures sections.
  Interventions: Other: Neuropsychological assessment
- Traumatic Brain Injury: Specific inclusion criteria for this participants' group are:
  * presence of a traumatic brain injury episode
  * absence of previous neurological and psychiatric conditions.
  There are no specific exclusion criteria for this participants' group (see general exclusion criteria).
  Participants will undergo a detailed neuropsychological assessment as detailed in the study's detailed description and outcome measures sections.
  Interventions: Other: Neuropsychological assessment
- Right Hemispheric Brain Tumor: Specific inclusion criteria for this participants' group are:
  - unilateral right hemispheric brain tumor.
  There are no specific exclusion criteria for this participants' group (see general exclusion criteria).
  Participants will undergo a detailed neuropsychological assessment as detailed in the study's detailed description and outcome measures sections.
  Interventions: Other: Neuropsychological assessment
- Left Hemispheric Brain Tumor: Specific inclusion criteria for this participants' group are:
  - unilateral left hemispheric brain tumor.
  There are no specific exclusion criteria for this participants' group (see general exclusion criteria).
  Participants will undergo a detailed neuropsychological assessment as detailed in the study's detailed description and outcome measures sections.
  Interventions: Other: Neuropsychological assessment
- Mild Cognitive Impairment: Specific inclusion criteria for this participants' group are:
  * MCI diagnosis according to Petersen et al., 2006 criteria
  * absence of previous neurological and psychiatric conditions.
  There are no specific exclusion criteria for this participants' group (see general exclusion criteria).
  Participants will undergo a detailed neuropsychological assessment as detailed in the study's detailed description and outcome measures sections.
  Interventions: Other: Neuropsychological assessment
- Healthy Individuals: Specific inclusion criteria for this participants' group are:
  - absence of neurological and psychiatric conditions.
  There are no specific exclusion criteria for this participants' group (see general exclusion criteria).
  Participants will undergo a detailed neuropsychological assessment as detailed in the study's detailed description and outcome measures sections.
  Interventions: Other: Neuropsychological assessment

INTERVENTIONS:
Other: Neuropsychological assessment — * APACS assessing various aspects of pragmatic communication abilities;
  * SET assessing cognitive and emotional theory of mind;
  * COAST assessing functional communication impairments in daily activities and their impact on the quality of life after the illness onset;
  * PWB assessing the individual's perceived quality of life and psychological well-being;
  * other neuropsychological assessment tools depending on the participant's pathology and routinely used in the clinical practice within the Institution.

SUMMARY:
Pragmatics of language refers to the set of abilities that allow one to use and interpret language according to context and, in general, to communicate effectively. Disorders in the pragmatics of language are prevalent in various clinical populations. They are a cause of social withdrawal and worse quality of life, both for patients directly affected and for their family members. Despite this, this type of disorder is rarely considered in neuropsychological assessment and rehabilitation.

This study's objective is to characterize pragmatic deficits in various neurological populations, allowing for the most accurate diagnosis possible and leading to the planning of personalized and effective Rehabilitation Plans.

DETAILED DESCRIPTION:
To delineate the pragmatic deficit profile for each pathology group, eligible participants will undergo a neuropsychological assessment, subdivided into as many sessions as per the participant's availability and tolerance.

Assessment tools will include:

* APACS (A test for the Assessment of Pragmatic Abilities and Cognitive Substrates; Arcara and Bambini, 2016)
* SET (Story-based Empathy Task, Dodich et al., 2015)
* COAST (Communication Outcome After Stroke, Bambini et al., 2016)
* PWB (Psychological Well-Being scales, Sirigatti et al., 2009)
* other neuropsychological assessment tools depending on the participant's pathology and routinely used in the clinical practice within the Institution.

Resulting test scores will be statistically analyze to provide pragmatic and cognitive profiles for each pathology.

ELIGIBILITY:
Inclusion Criteria:

* Presence of objective neuropsychological assessment using standardized tests used in clinical routine.
* Ability to knowingly provide written informed consent and , therefore preserved comprehension skills and good understanding of simple verbal requests (for the experimental phase).
* Being a native speaker of Italian.

Exclusion Criteria:

* Presence of disability that impairs participation in research.
* Insufficient knowledge of the Italian language.
* Refusal to participate in the research.
* Other relevant prior neurological or psychiatric conditions (other than those determining membership in the experimental group).
* Comorbidity of multiple conditions that would determine membership in more than one experimental group.
* Comorbidity with other neurological conditions.
* Presence of prior psychiatric conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurological patients and healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 324 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pragmatic Profile | after enrollmnet (T0)
  results at ASsessemnt of Pragmatics Abilities and Cognitive Substrates (APACS) test

SECONDARY OUTCOMES:
Theory of Mind | after enrollmnet (T0)
  Results at Story Empathy Test (SET) score
Functional Communication Abilities | after enrollmnet (T0)
  Results at Communication Outcome After Stroke (COAST)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Arcara, Principal Investigator — San Camillo IRCCS Hospital
Locations (1):
- San Camillo IRCCS s.r.l., Venice-Lido, Venice, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arcara G, Bambini V. A Test for the Assessment of Pragmatic Abilities and Cognitive Substrates (APACS): Normative Data and Psychometric Properties. Front Psychol. 2016 Feb 12;7:70. doi: 10.3389/fpsyg.2016.00070. eCollection 2016. PMID 26903894
- [Background] Bambini, V., Arcara, G., Aiachini, B., Cattani, B., Dichiarante, M. L., Moro, A., ... & Pistarini, C. (2017). Assessing functional communication: validation of the Italian versions of the Communication Outcome after Stroke (COAST) scales for speakers and caregivers. Aphasiology, 31(3), 332-358.
- [Background] Dodich A, Cerami C, Canessa N, Crespi C, Iannaccone S, Marcone A, Realmuto S, Lettieri G, Perani D, Cappa SF. A novel task assessing intention and emotion attribution: Italian standardization and normative data of the Story-based Empathy Task. Neurol Sci. 2015 Oct;36(10):1907-12. doi: 10.1007/s10072-015-2281-3. Epub 2015 Jun 14. PMID 26072203
- [Background] Sirigatti, S., Stefanile, C., Giannetti, E., Iani, L., Penzo, I., & Mazzeschi, A. (2009). Assessment of factor structure of Ryff's Psychological Well-Being Scales in Italian adolescents. Bollettino di Psicologia Applicata, 259(56), 30-50.